CLINICAL TRIAL: NCT06221618
Title: Evaluation of Vascular Structure in Elderly Using High-frequency Ultrasound and Construction of a Multimodal Risk Assessment System for Cardiovascular Diseases: a Multicenter Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Chinese PLA General Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Xuanwu Hospital, Beijing (Other); Shenzhen People's Hospital (Other); Shenzhen University (Other); The Fourth Affiliated Hospital of China Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202212(XZ)-015-1
Record Dates: First submitted 2023-12-18; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-12

CONDITIONS: Atherosclerosis; Stroke; Coronary Disease
Keywords: Stroke; Coronary heart disease; Risk assessment; Multimodality imaging; Cardiovascular diseases
MeSH Terms: conditions — Atherosclerosis; Stroke; Coronary Disease; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Coronary heart disease cohort: CCTA required for coronary heart disease cohort
  Interventions: Other: High-frequency carotid arteries ultrasound, CCTA, Cranial MRA
- Stroke cohort: Cranial MRA required for stroke cohort
  Interventions: Other: High-frequency carotid arteries ultrasound, CCTA, Cranial MRA
- Normal control group: Healthy elderly without coronary heart disease and stroke (≥ 60 years old)
  Interventions: Other: High-frequency carotid arteries ultrasound, CCTA, Cranial MRA

INTERVENTIONS:
Other: High-frequency carotid arteries ultrasound, CCTA, Cranial MRA — CCTA and carotid high-frequency ultrasound for all patients in the coronary heart disease cohort. Cranial MRA and carotid high-frequency ultrasound for all people in the stroke cohort.Carotid high-frequency ultrasound for all patients in the normal control group.All patients were treated optimally according to guidelines

SUMMARY:
Coronary heart disease(CHD), stroke, and hypertension are major diseases that seriously affect human health.Pathologic changes in the arteries involved in the above diseases mainly occur in the intimal or medial layer of the arteries. Among them, cardiovascular and cerebrovascular diseases (CHD and stroke) have become the top two causes of death worldwide, with elderly patients accounting for the vast majority. CHD is an important cause of death, and atherosclerosis (AS) is the main pathology underlying it.AS predominantly occurs in the intima layer, and the use of high-resolution imaging techniques to visualize anatomical changes in the intima-media layer of the arteries alone is valuable for the study of AS. Coronary computed tomographic angiography (CCTA) and intracranial vascular magnetic resonance angiography (MRA) can clearly visualize coronary and intracranial arterial lesions, measure luminal stenosis and other important information, and provide a basis for diagnosis, treatment and prognosis of the disease. By integrating CCTA/MRA/Ultrasound multimodal imaging technology, investigators aim to develop a non-invasive CHD and stroke intelligent screening and evaluation system, which is bound to have great clinical and social value.

This study is a national multi-center follow-up observational study, which is expected to collect and establish a database of clinical and imaging information of no less than 20,000 cases of elderly subjects. Some data is derived from the pre-established database (>12,000 cases) in cooperative research centers, while additional data will be collected from the newly established prospective follow-up database. Investigators performed noninvasive high-frequency ultrasound to detect arterial vascular structural changes, vascular dynamics and other indicators based on the existing database and the newly established imaging database to explore the characteristics of carotid atherosclerosis changes and ultrasound monitoring methods in the elderly. Finally, investigators integrated clinical and multimodal noninvasive imaging information to construct a noninvasive imaging-based intelligent risk assessment system for CHD and stroke.

Primary endpoint was the cardiovascular-complex endpoint event,including myocardial infarction, cardiovascular death, resuscitation with cardiac arrest, revascularization, and stroke. Secondary endpoint was vascular lesion progression, including increase of vascular intima thickness, increase of vascular media thickness, plaque progression, and increase of vascular stenosis. All enrolled patients were followed up every six months to record whether the primary endpoint and secondary endpoint events occurred and to record the time and type of occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* All patients had original ultrasound images of bilateral carotid arteries with DICOM format and arteriosclerosis clinical and laboratory data
* Original data of CCTA or examination results in the baseline status are needed for CHD patients
* Original data of intracranial artery MRA or examination results in the baseline status are needed for patients with ischemic stroke.

Exclusion Criteria:

* Age is <60 years old
* Severe cardiac insufficiency, New York Heart Association(NYHA) class IV and (or) left ventricular ejection fraction <30%
* Uncontrollable severe hypertension (systolic blood pressure≥ 180 mmHg or diastolic blood pressure≥ 110 mmHg) or uncontrollable severe diabetes mellitus, i.e., diabetes mellitus complicated with acute complications (including diabetic ketoacidosis and hypertonic hyperglycemic nonketosis coma), or acute hyperglycemic state (random blood glucose> 16.7mmol/L and (or) blood ketone 1.0-3.0mmol/L) without acute complications
* Severe valvular disease (moderate regurgitation and / or stenosis in each valve)
* Various cardiomyopathy caused by hypertrophic cardiomyopathy, dilated cardiomyopathy, alcoholic cardiomyopathy, myocardial amyloidosis
* Severe arrhythmia: persistent atrial fibrillation or atrial flutter, degree II 2 and above atrioventricular block, complete left bundle branch block
* Severe hepatic and renal insufficiency (glutamate transaminase and / or glutamine transaminase> 3 times the upper limit of normal value, Blood creatinine> 134 μmol/L or an estimated glomerular filtration rate of <60ml/min/1.73m2)
* Severe chronic obstructive pulmonary disease or asthma
* Severe non-cardiovascular disease (malignant tumor, thyroid disease, infection, connective tissue disease)
* Mental retardation or mental disorders
* Life expectancy <3 years due to various factors
* Refusal to sign informed consent
* Allergy to contrast agent should also be ruled out for patients undergoing CCTA for CHD.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients come from the following hospitals:
  * Qilu Hospital of Shandong University,
  * Xuanwu Hospital of Capital Medical University,
  * Chinese PLA General Hospital
  * Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
  * Shenzhen People's Hospital
  * The Fourth Affiliated Hospital of China Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular and cerebrovascular composite endpoint events | From the date of enrollment until the date of the first recorded endpoint event or the date of the end of the study, up to 20 months
  * Myocardial infarction
  * Cardiovascular death
  * Resuscitation with cardiac arrest
  * Revascularization
  * Stroke.

SECONDARY OUTCOMES:
Progression of the vascular lesions | From the date of enrollment until the date of the first recorded endpoint event or the date of the end of the study, up to 20 months
  * Increase of vascular intima thickness
  * Increase of vascular media thickness
  * Plaque progression
  * Increase of vascular stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Mei Zhang, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Mei Zhang, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lusis AJ. Atherosclerosis. Nature. 2000 Sep 14;407(6801):233-41. doi: 10.1038/35025203. PMID 11001066
- [Background] Schoenhagen P, Vince DG. Intravascular photoacoustic tomography of coronary atherosclerosis: riding the waves of light and sound. J Am Coll Cardiol. 2014 Jul 29;64(4):391-3. doi: 10.1016/j.jacc.2014.05.018. No abstract available. PMID 25060375
- [Background] Ruengsakulrach P, Sinclair R, Komeda M, Raman J, Gordon I, Buxton B. Comparative histopathology of radial artery versus internal thoracic artery and risk factors for development of intimal hyperplasia and atherosclerosis. Circulation. 1999 Nov 9;100(19 Suppl):II139-44. doi: 10.1161/01.cir.100.suppl_2.ii-139. PMID 10567293